CLINICAL TRIAL: NCT01633736
Title: Targeted Hip Progressive Resistance Training to Improve Single Leg Balance and Walking in Children With Cerebral Palsy
Brief Title: Targeted Hip Strength Training in Children With Cerebral Palsy (CP)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UoN-SWW-2
Record Dates: First submitted 2012-06-15; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Cerebral Palsy
Keywords: single blinded; randomised; controlled; physiotherapy; children; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- home progressive resistance exercise (Experimental)
  Interventions: Other: Usual care plus progresive resistance training

INTERVENTIONS:
Other: Usual care plus progresive resistance training — Duration 8 weeks; two weeks of familiarisation with the intervention protocol without resistance (for familiarisation and neural adaptation) followed by 6 weeks progressive resistance (PR). The three times a week PR training will be as a home exercise program with fortnightly home visits to monitor/progress PR training. It comprises a 4 minute warm up and cool down with one exercise targeting the hip abductors and one the lateral rotators. Exercise prescription will follow existing guidelines for progressive PR training. Parents will be taught supervision by the researcher using clear explanations in words and pictures in a logbook. Logbooks have been found to facilitate compliance, dosage and motivation.
  Other Names: strength training

SUMMARY:
This study's main aim is to look at targeted strength training for muscles at the hips. Specifically to consider whether targeted strength training not only effects strength of the specific muscles but also ability to stand on one leg (single leg balance) as well as walking in children with cerebral palsy? This study is a feasibility of method of investigation.

DETAILED DESCRIPTION:
This study is focusing on functional change. The reasoning is that if the targeted strength training is effective at improving hip muscle contribution to stability then single leg balance may be improved. This may be functionally evident when weight bearing is taken by say the left leg in gait (percentage stance phase of gait) and as a consequence the opposing swing phase will be optimised as measured by stride. Thus the research question is does strengthening of the rotating and sideways moving hip muscles improve the walking of children with CP as measured by appropriate aspects of gait? Secondly, does this targeted strengthening also increase duration of single leg balance which is a simple easy to use measure in the community without the need for specialised equipment? The primary outcome measure will use a laboratory based 4 camera Codsmotion (CODA) biomechanical analysis system to measure stride (a) and percentage duration of stance phase of gait (b). Secondarily the duration of single leg balance in terms of seconds will be recorded. Gross motor functional and quality of life as also being assessed. The intervention is strengthening which will be implemented with the principles of progressive resistance training. Children with CP's therapists would ask for this type of intervention to be carried out

ELIGIBILITY:
Inclusion Criteria:

* Children with CP aged between 7-16 years having sufficient cognition to undertake a strength training program

Exclusion Criteria:

1. non-ambulation children or those unable to walk 5 meters independently (without walking aid),
2. lower limb surgery within 12 months,
3. botox within 6 months,
4. oral muscle relaxant medication
5. significant learning difficulty
6. Any concurrent condition which would be contraindicated to progressive resistance training such as unmanaged high blood pressure, cardiac pathology or uncontrolled epilepsy
7. Where at baseline assessment finds no weakness in the muscles under investigation
8. concurrent or within 6 months involvement in any other research study
9. Non consent to General Practitioner (GP) notification.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Gait parameter | baseline, plus 8 weeks and plus 8 weeks (exit point)
  4 camera CODA gait analysis system for change in percentage stance phase of gait and stride in cm.

SECONDARY OUTCOMES:
Gross Motor Function Measure (GMFM) | Baseline, plus 8 weeks and plus 8 weeks (exit)
  To investigate any change in dimensions D and E of fucntioal activity with standardised GMFM.

CONTACTS AND LOCATIONS:
Overall Officials: Grahame Pope, MPhil, BSc, Principal Investigator — The University of Nottingham
Locations (1):
- Divison of Physiotherapy, School of Nursing, Midwifery and Physiotherapy, The University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Cans, C., et al., Recommendations from the SCPE collaborative group for defining and classifying cerebral palsy. , in The Definition and Classification of Cerebral Palsy, P. Baxter, Editor. 2003, the SCPE collaborative group.
- [Background] Reddihough DS, Collins KJ. The epidemiology and causes of cerebral palsy. Aust J Physiother. 2003;49(1):7-12. doi: 10.1016/s0004-9514(14)60183-5. PMID 12600249
- [Background] Hemming K, Hutton JL, Pharoah PO. Long-term survival for a cohort of adults with cerebral palsy. Dev Med Child Neurol. 2006 Feb;48(2):90-5. doi: 10.1017/S0012162206000211. PMID 16417662
- [Background] Koman LA, Smith BP, Shilt JS. Cerebral palsy. Lancet. 2004 May 15;363(9421):1619-31. doi: 10.1016/S0140-6736(04)16207-7. PMID 15145637
- [Background] Krigger KW. Cerebral palsy: an overview. Am Fam Physician. 2006 Jan 1;73(1):91-100. PMID 16417071
- [Background] Parkes J, Donnelly M, Dolk H, Hill N. Use of physiotherapy and alternatives by children with cerebral palsy: a population study. Child Care Health Dev. 2002 Nov;28(6):469-77. doi: 10.1046/j.1365-2214.2002.00304.x. PMID 12568476
- [Background] Himpens E, Van den Broeck C, Oostra A, Calders P, Vanhaesebrouck P. Prevalence, type, distribution, and severity of cerebral palsy in relation to gestational age: a meta-analytic review. Dev Med Child Neurol. 2008 May;50(5):334-40. doi: 10.1111/j.1469-8749.2008.02047.x. Epub 2008 Mar 18. PMID 18355333
- [Background] Pallant, J (2001) SPSS Survival Manual. Edition 10, Open University Press, Buckingham.Philadelphia
- [Background] Elder GC, Kirk J, Stewart G, Cook K, Weir D, Marshall A, Leahey L. Contributing factors to muscle weakness in children with cerebral palsy. Dev Med Child Neurol. 2003 Aug;45(8):542-50. doi: 10.1017/s0012162203000999. PMID 12882533
- [Background] Levitt, S., Treatment of Cerebral Palsy and Motor Delay. 3rd Edition ed. 1995: Blackwell Science.
- [Background] Ross SA, Engsberg JR. Relation between spasticity and strength in individuals with spastic diplegic cerebral palsy. Dev Med Child Neurol. 2002 Mar;44(3):148-57. doi: 10.1017/s0012162201001852. PMID 12005315
- [Background] Scholtes VA, Dallmeijer AJ, Rameckers EA, Verschuren O, Tempelaars E, Hensen M, Becher JG. Lower limb strength training in children with cerebral palsy--a randomized controlled trial protocol for functional strength training based on progressive resistance exercise principles. BMC Pediatr. 2008 Oct 8;8:41. doi: 10.1186/1471-2431-8-41. PMID 18842125
- [Background] Wiley ME, Damiano DL. Lower-extremity strength profiles in spastic cerebral palsy. Dev Med Child Neurol. 1998 Feb;40(2):100-7. doi: 10.1111/j.1469-8749.1998.tb15369.x. PMID 9489498
- [Background] Damiano DL, Kelly LE, Vaughn CL. Effects of quadriceps femoris muscle strengthening on crouch gait in children with spastic diplegia. Phys Ther. 1995 Aug;75(8):658-67; discussion 668-71. doi: 10.1093/ptj/75.8.658. PMID 7644570
- [Background] Tran, Q.T., Cerebral palsy; considerations for training. Strength and Conditioning Journal, 2005. 27(6): p. 34-38
- [Background] Damiano DL, Dodd K, Taylor NF. Should we be testing and training muscle strength in cerebral palsy? Dev Med Child Neurol. 2002 Jan;44(1):68-72. doi: 10.1017/s0012162201001682. No abstract available. PMID 11811654
- [Background] Dodd KJ, Taylor NF, Damiano DL. A systematic review of the effectiveness of strength-training programs for people with cerebral palsy. Arch Phys Med Rehabil. 2002 Aug;83(8):1157-64. doi: 10.1053/apmr.2002.34286. PMID 12161840
- [Background] Pippenger WS, Scalzitti DA. What are the effects, if any, of lower-extremity strength training on gait in children with cerebral palsy? Phys Ther. 2004 Sep;84(9):849-58. No abstract available. PMID 15330697
- [Background] Morton JF, Brownlee M, McFadyen AK. The effects of progressive resistance training for children with cerebral palsy. Clin Rehabil. 2005 May;19(3):283-9. doi: 10.1191/0269215505cr804oa. PMID 15859529
- [Background] Lee JH, Sung IY, Yoo JY. Therapeutic effects of strengthening exercise on gait function of cerebral palsy. Disabil Rehabil. 2008;30(19):1439-44. doi: 10.1080/09638280701618943. PMID 19230216
- [Background] Fowler EG, Ho TW, Nwigwe AI, Dorey FJ. The effect of quadriceps femoris muscle strengthening exercises on spasticity in children with cerebral palsy. Phys Ther. 2001 Jun;81(6):1215-23. PMID 11380277
- [Background] Blundell SW, Shepherd RB, Dean CM, Adams RD, Cahill BM. Functional strength training in cerebral palsy: a pilot study of a group circuit training class for children aged 4-8 years. Clin Rehabil. 2003 Feb;17(1):48-57. doi: 10.1191/0269215503cr584oa. PMID 12617379
- [Background] Damiano DL, Abel MF. Functional outcomes of strength training in spastic cerebral palsy. Arch Phys Med Rehabil. 1998 Feb;79(2):119-25. doi: 10.1016/s0003-9993(98)90287-8. PMID 9473991
- [Background] Seniorou M, Thompson N, Harrington M, Theologis T. Recovery of muscle strength following multi-level orthopaedic surgery in diplegic cerebral palsy. Gait Posture. 2007 Oct;26(4):475-81. doi: 10.1016/j.gaitpost.2007.07.008. Epub 2007 Sep 12. PMID 17855096
- [Background] Johnson, L.M., et al., The effect of plantarflexor muscle strengthening on the gait and range of motion at the ankle in ambulant children with cerebral palsy: a pilot study. New Zealand Journal of Physiotherapy, 1998. April: p. 8-14.
- [Background] Engsberg JR, Ross SA, Collins DR. Increasing ankle strength to improve gait and function in children with cerebral palsy: a pilot study. Pediatr Phys Ther. 2006 Winter;18(4):266-75. doi: 10.1097/01.pep.0000233023.33383.2b. PMID 17108800
- [Background] Unnithan VB, Katsimanis G, Evangelinou C, Kosmas C, Kandrali I, Kellis E. Effect of strength and aerobic training in children with cerebral palsy. Med Sci Sports Exerc. 2007 Nov;39(11):1902-9. doi: 10.1249/mss.0b013e3181453694. PMID 17986896
- [Background] Perry, J., Gait Analysis Normal and Pathological Function. 1992, Thorofare, NJ: SLACK Inc. 502.
- [Background] Gage JR, Novacheck TF. An update on the treatment of gait problems in cerebral palsy. J Pediatr Orthop B. 2001 Oct;10(4):265-74. PMID 11727367
- [Background] Palastanga, N., D. Field, and R. Soames, Anatomy and Human Movement structure and function Vol. 5th. 2006: Elsevier.
- [Background] Darrah, J., et al., Review of the effects of progressive resisted muscle strengthening in children with cerebral palsy: a clinical consensus exercise. Pediatric Physical Therapy, 1997. 9: p. 12-17.
- [Background] Anttila H, Autti-Ramo I, Suoranta J, Makela M, Malmivaara A. Effectiveness of physical therapy interventions for children with cerebral palsy: a systematic review. BMC Pediatr. 2008 Apr 24;8:14. doi: 10.1186/1471-2431-8-14. PMID 18435840
- [Background] Verschuren O, Ketelaar M, Takken T, Helders PJ, Gorter JW. Exercise programs for children with cerebral palsy: a systematic review of the literature. Am J Phys Med Rehabil. 2008 May;87(5):404-17. doi: 10.1097/PHM.0b013e31815b2675. PMID 17993987
- [Background] Armstrong, N. and W. van Mechelen, Paediatric exercise science and medicine. 2nd ed. 2008: Oxford University Press
- [Background] American Academy of Pediatrics Committee on Sports Medicine: Strength training, weight and power lifting, and body building by children and adolescents. Pediatrics. 1990 Nov;86(5):801-3. No abstract available. PMID 2235239
- [Background] Liao HF, Liu YC, Liu WY, Lin YT. Effectiveness of loaded sit-to-stand resistance exercise for children with mild spastic diplegia: a randomized clinical trial. Arch Phys Med Rehabil. 2007 Jan;88(1):25-31. doi: 10.1016/j.apmr.2006.10.006. PMID 17207671
- [Background] Patikas D, Wolf SI, Mund K, Armbrust P, Schuster W, Doderlein L. Effects of a postoperative strength-training program on the walking ability of children with cerebral palsy: a randomized controlled trial. Arch Phys Med Rehabil. 2006 May;87(5):619-26. doi: 10.1016/j.apmr.2006.01.023. PMID 16635623
- [Background] Brooks, G., Fahey. TD., and K. Baldwin, Exercise physiology; human bioenergetics and its applications. 4th ed. 2004: McGraw Hill.
- [Background] Behm DG, Faigenbaum AD, Falk B, Klentrou P. Canadian Society for Exercise Physiology position paper: resistance training in children and adolescents. Appl Physiol Nutr Metab. 2008 Jun;33(3):547-61. doi: 10.1139/H08-020. PMID 18461111
- [Background] Patikas D, Wolf SI, Armbrust P, Mund K, Schuster W, Dreher T, Doderlein L. Effects of a postoperative resistive exercise program on the knee extension and flexion torque in children with cerebral palsy: a randomized clinical trial. Arch Phys Med Rehabil. 2006 Sep;87(9):1161-9. doi: 10.1016/j.apmr.2006.05.014. PMID 16935049
- [Background] Verschuren O, Ketelaar M, Gorter JW, Helders PJ, Uiterwaal CS, Takken T. Exercise training program in children and adolescents with cerebral palsy: a randomized controlled trial. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1075-81. doi: 10.1001/archpedi.161.11.1075. PMID 17984410
- [Background] van der Linden ML, Aitchison AM, Hazlewood ME, Hillman SJ, Robb JE. Test-Retest repeatability of gluteus maximus strength testing using a fixed digital dynamometer in children with cerebral palsy. Arch Phys Med Rehabil. 2004 Dec;85(12):2058-63. doi: 10.1016/j.apmr.2003.12.037. PMID 15605348
- [Background] van den Beld WA, van der Sanden GA, Sengers RC, Verbeek AL, Gabreels FJ. Validity and reproducibility of hand-held dynamometry in children aged 4-11 years. J Rehabil Med. 2006 Jan;38(1):57-64. doi: 10.1080/16501970510044043. PMID 16548089
- [Background] Varni JW, Burwinkle TM, Berrin SJ, Sherman SA, Artavia K, Malcarne VL, Chambers HG. The PedsQL in pediatric cerebral palsy: reliability, validity, and sensitivity of the Generic Core Scales and Cerebral Palsy Module. Dev Med Child Neurol. 2006 Jun;48(6):442-9. doi: 10.1017/S001216220600096X. PMID 16700934
- [Background] Coe R (2002) It's the Effect Size, Stupid; What effect size is and why it is important Paper presented at the Annual Conference of the British Educational Research Association, University of Exeter, England, 12-14 September 2002